CLINICAL TRIAL: NCT03168100
Title: University of Arkansas (UARK# 2017-03): A Single-Arm, Open-label Study of Anti-SLAMF7 mAb Therapy After Autologous Stem Cell Transplant in Patients With Multiple Myeloma (Total Therapy 8)
Brief Title: 2017-03: A Single-Arm, Open-label Study of Anti-Signaling Lymphocytic Activation Molecule F7 (Anti-SLAMF7) Monoclonal Antibody (mAb) Therapy After Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No study population. No subjects enrolled.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206603
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Treatment (Experimental): Elotuzumab (10 mg Days 1 and 15), lenalidomide (15 mg Days 1-21), and dexamethasone (20 mg days 1, 8, 15, and 22) administered in 28-day cycles which will be alternated every 8 weeks with bortezomib (1.0 mg Days 1, 8, and 15), lenalidomide (15 mg Days 1-21), and dexamethasone (20 mg Days 1, 8, 15, and 22)
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Elotuzumab — administered via IV infusion
  Other Names: Empliciti
Drug: Lenalidomide — taken by mouth
  Other Names: Revlimid
Drug: Dexamethasone — taken by mouth
  Other Names: Decadron
Drug: Bortezomib — administered as a subcutaneous injection
  Other Names: Velcade

SUMMARY:
The Total Therapy treatment regimens developed at the Myeloma Institute have demonstrated great improvement in treatment outcomes for multiple myeloma patients. However, some patients still relapse early during maintenance treatment meaning that better options are still needed. This study will evaluate a treatment regimen that alternates two different 3-drug regimens every eight weeks for patients that have previously completed autologous stem cell transplant. The two regimens are bortezomib, lenalidomide, and dexamethasone (VRD) which will be alternated with Elotuzumab, lenalidomide, and dexamethasone (Elo RD). Effectiveness will be measured by the depth of response (i.e., whether or not minimal residual disease (MRD) negative status is achieved). The rate of MRD negativity from this study will be compared to historical control data from the Total Therapy 4 trial which used continuous VRD maintenance therapy after stem cell transplant(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age and not older than 75 years of age at the time of enrollment.
* Patients must have completed a stem cell transplant regimen for newly diagnosed multiple myeloma (MM) consisting of (at least) induction chemotherapy and single or tandem autologous stem cell transplant (ASCT) within eight months of study enrollment. The completed regimen may have included post-transplant consolidation therapy, but post-transplant consolidation is not required.
* Patients must have achieved at least a partial response (PR) (according to International Myeloma Working Group (IMWG) criteria) in response to the completed transplant regimen.
* ECOG ≤ 2 (ECOG of 3 allowed if solely due to symptoms of MM-related bone disease).
* Patients must have absolute neutrophil count (ANC) ≥ 1,000/mm3 and a platelet count of ≥ 75,000/μL.
* Patients must have a baseline serum creatinine level of < 3 mg/dL and baseline alanine aminotransferase (ALT) < 3x Upper limit of normal (ULN)
* Toxicities related to prior therapies must be resolved to ≤ Grade 2 according to NCI Common Terminology for Adverse Events (CTCAE) Version 4.
* Female patients must be:

  * Postmenopausal for at least 1 year before the screening visit, OR
  * Surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 simultaneous effective methods of contraception, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, post-vasectomy) must agree to one of the following:

  * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must sign an Institutional Review Board (IRB)-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* Female patients who are nursing or pregnant may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of beginning study treatment. Refer to the Revlimid Risk Evaluation and Mitigation Strategies (REMS) program for more information.
* History of poorly controlled hypertension, diabetes mellitus, active or uncontrolled hepatitis, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol, or that in the opinion of the investigator would constitute a hazard for participating in this study.
* History of clinically significant cardiac disease as determined by the enrolling physician including cardiac amyloidosis.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will be acceptable if the patient's life expectancy exceeds five years.
* Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins or any of the study medications, their analogues, or excipients in the various formulations of any agent (refer to the latest versions of the package inserts).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Depth of Response | Six months from start of study treatment.
  Depth of response will be measured by minimal residual disease (MRD) status (i.e., positive or negative).

CONTACTS AND LOCATIONS:
Overall Officials: Faith Davies, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.